CLINICAL TRIAL: NCT03329638
Title: A Phase II, Randomized, Double-Masked, Placebo-Controlled, Parallel-Group Study Assessing the Efficacy and Safety of DE-127 Ophthalmic Solution Compared With Placebo in Subjects With Mild or Moderate Myopia (APPLE)
Brief Title: A Study Assessing the Efficacy and Safety of DE-127 Ophthalmic Solution in Subjects With Mild or Moderate Myopia (APPLE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012701LT
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DE-127 Ophthalmic Solution low dose (Experimental)
  Interventions: Drug: DE-127 Ophthalmic Solution low dose
- DE-127 Ophthalmic Solution medium dose (Experimental)
  Interventions: Drug: DE-127 Ophthalmic Solution medium dose
- DE-127 Ophthalmic Solution high dose (Experimental)
  Interventions: Drug: DE-127 Ophthalmic Solution high dose
- Placebo Ophthalmic Solution (Placebo Comparator)
  Interventions: Drug: Placebo Ophthalmic Solution

INTERVENTIONS:
Drug: DE-127 Ophthalmic Solution low dose — Low dose of DE-127 Ophthalmic Solution dosed once daily for 12 months
  Arms: DE-127 Ophthalmic Solution low dose
Drug: DE-127 Ophthalmic Solution medium dose — Medium dose of DE-127 Ophthalmic Solution dosed once daily for 12 months
  Arms: DE-127 Ophthalmic Solution medium dose
Drug: DE-127 Ophthalmic Solution high dose — High dose of DE-127 Ophthalmic Solution dosed once daily for 12 months
  Arms: DE-127 Ophthalmic Solution high dose
Drug: Placebo Ophthalmic Solution — Placebo Ophthalmic Solution dosed once daily for 12 months
  Arms: Placebo Ophthalmic Solution

SUMMARY:
To investigate the safety and efficacy of three concentrations of DE-127 ophthalmic solution when compared to Placebo in subjects diagnosed with mild or moderate myopia.

To investigate the dose response of DE-127.

ELIGIBILITY:
Inclusion Criteria:

* Refractive error of spherical equivalent -1.0 diopter to -6.0 diopter in both eyes
* Anisometropia of spherical equivalent less than or equal to 1.50 diopter in both eyes
* Distance vision correctable to logMAR 0.2 or better in both eyes
* Normal intraocular pressure of not greater than 21 mmHg in both eyes
* No allergy to atropine, cyclopentolate, proparacaine and benzalkonium chloride

Exclusion Criteria:

* Amblyopia or manifest strabismus including intermittent tropia
* Ocular disorders that potentially affect myopia or refractive power
* Previous or current use of contact lenses, bifocal lenses, progressive addition lenses, or other forms of treatment (including atropine and pirenzepine) for myopia
* Systemic disorders that potentially affect myopia or refractive power

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
Spherical equivalent | Month 12
  Change from Baseline in spherical equivalent determined by cycloplegic autorefraction at Month 12 in the study eye.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore